CLINICAL TRIAL: NCT05032807
Title: Pharmacokinetic Study of a Novel Lipid Formulation of Cannabidiol Compared to a Standard Formulation
Acronym: CLIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS: 288415
Record Dates: First submitted 2021-08-25; First posted 2021-09-02 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Absorption; Chemicals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel lipid formulation then standard formulation (Experimental)
  Interventions: Drug: Standard formulation; Drug: Novel formulation
- Standard formulation then lipid formulation (Experimental)
  Interventions: Drug: Standard formulation; Drug: Novel formulation

INTERVENTIONS:
Drug: Standard formulation — Cannabidiol 1000mg standard formulation, single dose, oral
Drug: Novel formulation — Cannabidiol 1000mg with lipid matrix, single dose, oral

SUMMARY:
Cannabidiol (CBD) has been approved as a treatment for rare childhood epilepsies and could be an effective treatment for psychotic disorders, anxiety disorders and addictions. It is available as an oral liquid and as standard oral capsules.

The bioavailability of oral cannabidiol is poor (only around 5-10% is absorbed), particularly in the fasted state. With food, its absorption is much higher. In one study, a high-fat breakfast increased the maximum plasma concentration by 4-5 times. As a result of this food effect, when prescribing standard oral formulations of CBD, clinicians should provide advice on dosing the drug according to mealtimes, otherwise, there may be an increased risk of side effects or limited effectiveness.

One way to reduce the food effect and improve bioavailability is to use lipid excipients. In the present study, the investigators will evaluate CBD at the dose that is effective in patients with chronic psychosis (1000mg). The novel formulation will use lipids that are all EU pharmacopoeia approved and have been used in medicinal products before.

The study aims to assess whether a novel lipid formulation can increase the bioavailability of oral CBD in the fasting state.

ELIGIBILITY:
Inclusion criteria i. Healthy volunteers. Defined as healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine.

ii. Age 18-45 iii. Agreeing to fast 15 hours; 10pm-1pm on dosing days iv. Capable of giving informed consent v. Written informed consent from participant

Exclusion criteria i. Clinically relevant medical history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the participant.

ii. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.

iii. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any neurological or mental illness.

iv. Surgery or medical condition that might affect absorption of medicines. v. Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min. Repeat measurements are permitted if values are borderline (i.e. values that are within 5 mm Hg for blood pressure or 5 beats/min for heart rate) or if requested by the investigator. Subjects can be included if the repeat value is within range or still borderline but deemed not clinically significant by the investigator.

vi. Loss of more than 400 mL blood during the 3 months before the trial, e.g. as a blood donor.

vii. Any prescribed medication (apart from contraceptives) viii. Use of any CBD products within six months of IMP administration ix. Use of any over-the-counter medications or health supplements within the past 2 weeks x. BMI <18 or >30.0kg/m2 xi. History of alcohol or substance misuse disorder xii. Intake of more than 14 units of alcohol weekly. xiii. Smokes more than 10 cigarettes per day xiv. Use of any illicit substances within the last six months of IMP administration xv. Pregnant or breastfeeding xvi. Women of childbearing potential (as defined in CTFG guidelines, see 5.7 Concomitant Medication) not willing to use a highly effective form of contraception (as defined in CTFG guidelines, see section 5.7 Concomitant Medication) during participation in the study or male patients not willing to ensure use of a condom during participation in the study.

xvii. eGFR≤ 70 mls/min xviii. Any liver function or renal function test abnormality. A repeat is allowed on one occasion for determination of eligibility.

xix. Urine drug screen positive for any substances xx. Positive alcohol breath test xxi. Participant in any other clinical trial or experimental drug study in the past 3 months xxii. Known hypersensitivity to CBD and/or SEEK formulation excipients xxiii. Participant is not able to swallow capsules

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chesney E, Mazibuko N, Oliver D, Minichino A, Lamper AD, Chester L, Reilly TJ, Lloyd M, Krakstrom M, Dickens AM, Oresic M, Lynch E, Stoloff G, Mehta MA, McGuire P. Novel Lipid Formulation Increases Absorption of Oral Cannabidiol (CBD). Pharmaceutics. 2024 Dec 1;16(12):1537. doi: 10.3390/pharmaceutics16121537. PMID 39771516

RESULTS

PARTICIPANT FLOW:
Groups:
- Novel Lipid Formulation Cannabidiol, Then Standard Formulation Cannabidiol: Cannabidiol novel formulation: Cannabidiol 1000mg with lipid matrix, single dose, oral
  Cannabidiol standard formulation: Cannabidiol 1000mg, single dose, oral
- Standard Formulation Cannabidiol, Then Novel Lipid Formulation Cannabidiol: Cannabidiol standard formulation: Cannabidiol 1000mg, single dose, oral
  Cannabidiol novel formulation: Cannabidiol 1000mg with lipid matrix, single dose, oral
Period: Treatment 1
Arm/Group | Novel Lipid Formulation Cannabidiol, Then Standard Formulation Cannabidiol | Standard Formulation Cannabidiol, Then Novel Lipid Formulation Cannabidiol
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Novel Lipid Formulation Cannabidiol, Then Standard Formulation Cannabidiol | Standard Formulation Cannabidiol, Then Novel Lipid Formulation Cannabidiol
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Novel Lipid Formulation Then Standard Formulation: Period 1: Cannabidiol 1000mg with lipid matrix, single dose, oral
  Period 2: Cannabidiol standard formulation: Cannabidiol 1000mg standard formulation, single dose, oral
- Standard Formulation Then Novel Lipid Formulation: Period 1: Cannabidiol standard formulation: Cannabidiol 1000mg standard formulation, single dose, oral
  Period 2: Cannabidiol novel formulation: Cannabidiol 1000mg with lipid matrix, single dose, oral
- Total: Total of all reporting groups
Arm/Group | Novel Lipid Formulation Then Standard Formulation | Standard Formulation Then Novel Lipid Formulation | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (4.4) | 26.7 (5.1) | 26.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 9
  Asian | 3 | 1 | 4
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Drug Exposure. (Area Under the Curve to Infinity [AUC(Inf)]
Description: Difference in AUC(inf) for a single dose of oral CBD between the novel and standard formulations in the fasting state.
Time Frame: 0 - 48 hours
Population: AUCinf could not be calculated for three participants in the standard CBD arm as plasma levels were not falling at the final time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/ml
Groups:
- Novel Lipid Formulation Cannabidiol: Cannabidiol novel formulation: Cannabidiol 1000mg with lipid matrix, single dose, oral
- Standard Formulation Cannabidiol: Cannabidiol standard formulation: Cannabidiol 1000mg standard formulation, single dose, oral
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
Number analyzed (Participants) | 14 | 11
ng*h/ml | 674.9 (103.05) | 134.76 (88.70)

2. Secondary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: 0 - 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
Number analyzed (Participants) | 14 | 14
ng/ml | 73.00 (149.82) | 3.11 (103.55)

3. Secondary Outcome: Tmax
Description: Time after administration of drug when maximum plasma concentration is reached
Time Frame: 0 - 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
Number analyzed (Participants) | 14 | 14
hours | 4 [2 to 8] | 6 [3 to 48]

4. Secondary Outcome: Plasma Half-life (t½)
Description: Half-life
Time Frame: 0 - 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
Number analyzed (Participants) | 14 | 11
hours | 13.71 (5.89) | 51.83 (57.61)

5. Secondary Outcome: 48 Hour Drug Exposure (AUC0-48)
Description: Area under the concentration-time curve from time zero to 48hours
Time Frame: 0 - 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/ml
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
Number analyzed (Participants) | 14 | 14
ng*h/ml | 611.42 (104.60) | 66.79 (50.65)

6. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS) - Total Score
Description: The GSRS was used to assess gastrointestinal symptoms over the past 24 hours only. It is a 15-item rating scale, where each item is assessed with a 7-point Likert scale, scored from 1 to 7, and with higher scores indicating more severe symptoms. The total score is the mean score across items (minimum score=1; maximum sore=7).
Time Frame: The scale will be used pre-dose and at 24 and 48 hours post dose.
Measure: Mean (Standard Deviation); unit: Mean score
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
Number analyzed (Participants) | 14 | 14
Mean score
  Baseline/pre-dose | 1.09 (0.17) | 1.06 (0.09)
  24 hours post dose | 1.25 (0.36) | 1.06 (0.11)
  48 hours post dose | 1.09 (0.18) | 1.02 (0.04)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Novel Lipid Formulation Cannabidiol | Standard Formulation Cannabidiol
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 11/14 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Novel Lipid Formulation Cannabidiol (N=14) | Standard Formulation Cannabidiol (N=14)
Anxiety (Psychiatric disorders) | 1 | 0
Somnolence (Psychiatric disorders) | 7 | 2
Dizziness (Nervous system disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Other (General disorders) | 3 | 6

LIMITATIONS AND CAVEATS:
Halflife and AUCinf could not be calculated for all participants in the standard CBD arm as plasma levels were not falling at the final time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT05032807/Prot_001.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT05032807/SAP_000.pdf